CLINICAL TRIAL: NCT00058786
Title: Treatment of Chronic Lymphocytic B-Leukemia (B-CLL) With Human IL-2 Gene Modified and Human CD40 Ligand-Expressing Autologous Tumor Cells
Brief Title: Treatment of Chronic Lymphocytic B-Leukemia With IL-2 and CD-40 Autologous Tumor Cells
Acronym: CLIMAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Director/Professor, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11541; Climat; NCT00609076 (obsolete NCT alias)
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Lymphocytic B-Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Injection of IL-2-secreting CD40L-expressing autologous B-CLL cells — Patients may be treated with a minimum of three up to six injections of their IL-2-secreting and CD40L-expressing autologous B-CLL cells, separated by one to two weeks in an immunological treatment window, i.e. in the absence of concurrent cytotoxic therapy. Any patient whose disease regresses after the administration of 6 injections may be offered further injections (i.e. more than 6 injections) of tumor vaccine at the dose level previously administered, if enough vaccines are available. Patients will receive a fixed dose of IL-2 secreting B-CLL cells throughout the entire treatment protocol (see Section 5.8), determined by previous studies in acute leukemia and in neuroblastoma, in which this level of IL-2 production has been safe. The dose escalation of CD40L-expressing cells is designed to reach the IL2/CD40L ratio shown to be effective in our preclinical models of neuroblastoma and lymphoma.

SUMMARY:
This is a research study to determine the safety and dosage of special cells that may make the patients own immune system fight the cancer. To do this, we will put a special gene into cancer cells that have been taken from the patient. This will be done in the laboratory. This gene will make the cells produce interleukin 2 (IL-2), which is a natural substance that may help the immune system kill cancer cells. Additionally, we will stimulate the cancer cells with another natural protein called CD40 ligand (CD40L), which preclinical human and animal studies suggest will help IL-2 perform better. Some of these cells will then be put back into the body. The cells are grown with normal embryonic fibroblasts. Studies of cancers in animals and in cancer cells that are grown in laboratories suggest that combining substances like IL-2 and CD40L helps the body kill cancer cells.

The purpose of this study is to learn the side effects and the safest effective dose of these special cells on the disease

DETAILED DESCRIPTION:
Before starting treatment some of the cancer cells will be taken from the patient and separated in the laboratory. A specially produced human virus (adenovirus) that carries the IL-2 gene will be put into the cells. The rest of the cancer cells will be stimulated to express on their surface a substance called the human CD40 ligand. These substances (IL-2 and CD40L), already naturally present in the body, are meant to help the immune system fight the cancer.

In this study, the modified cancer cells will be injected under the skin. There will be up to six shots. We do not know the best amount of special cells to use, so different patients will get different numbers of cells.

After the first three shots (if more modified cancer cells are available), patients may be able to have three additional shots. After they have received six shots, they may be able to have additional shots if the cancer has gotten smaller and more of the cells are available.

A complete history and physical examination is necessary before a patient can be enrolled in the study. A physical examination will also be performed weekly for ten weeks after the injection, then on week twelve, then monthly for one year. Patients will then have yearly checkups for the next fifteen years. After the first and second shots, we will remove some of the modified cells that have been injected under the skin, to study them. We will do this by removing a section of skin (referred to as a skin biopsy) at the place where the cells were injected. These tests will help us to see whether or not the modified cells are killing cancer cells and whether or not the cancer cells are growing. If we suspect the cancer cells are growing, we may repeat this procedure after the third and fourth shots.

To study how the immunity is working in the patients system, we will take blood samples before the first injection, then weekly for 10 weeks, on week 12, once a month for a year, and then eventually once a year for fifteen years. These blood samples must be taken at The Methodist Hospital. The total amount of blood that will be obtained is approximately two to three tablespoonfuls, which is considered a safe amount. If the patient has additional injections, blood will be drawn prior to each injection. Additional office visits may be necessary.

If the patient decides to withdraw at any time during the study both samples and data collected during the study will be maintained with identifiers for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for administration of their vaccine if they present with B-CLL (not in Richter's transformation) with (group A) or without (group B) measurable disease. Untreated or complete remission patients will be enrolled for vaccine administration in a therapeutic (i.e. no chemotherapy) window of three months. If during these three months (necessary to complete the vaccine study) the patient presents with rapid clinical progression, he or she will be excluded from our current study and will receive treatment according to the standard institutional guidelines. IMPORTANT NOTE: Vaccine production for complete remission patients can only be achieved if tumor cells have been collected BEFORE entering complete remission.
* Patients must have a life expectancy of at least 10 weeks.
* Patients must have ECOG performance status of 0-2.
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and must have an absolute neutrophil count of >/= 500/uL, absolute lymphocyte count >/= 200/uL, hemoglobin >/= 8g/dL and platelet count >/= 50,000/uL.
* Patients must not be infected at time of protocol entry, and should not be receiving antibiotics (other than prophylactic trimethoprim sulfamethoxazole).
* Patients must be HIV-negative.
* Patients must be willing to practice appropriate birth control methods during the study and for 3 months after the study is concluded.
* Patients must not be suffering from an autoimmune disease (including active graft-versus-host disease-GvHD, refractory immune thrombocytopenia-ITP or refractory autoimmune hemolytic anemia-AIHA) and should not be receiving immunosuppressive drugs.
* Patients must have adequate liver function (total bilirubin </= 1.5mg/dl, SGOT </= 2 times normal, normal prothrombin time).
* Patients must have adequate renal function (creatinine < 3 times normal for age or creatinine clearance > 80mg/min/1.73m2).
* Patients must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side-effects. Patients will be given a copy of the consent form.
* Patient must not have received treatment with other investigational agents within the last 4 weeks.

Exclusion Criteria:

* Richter's transformation (aggressive non-Hodgkin's lymphoma)
* active infection
* significant autoimmune disease (including active GvHD, ITP and AIHA)
* requirement for immunosuppressive drugs
* inadequate liver and/or renal function
* pregnancy or lactation
* refusal to practice birth control methods
* seropositive for HIV
* life expectancy less than 10 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety of 3-6 SQ injections of autologous malignant B cells from chronic B-CLL pts, which have been modified ex vivo to secrete human interleukin-2 (hIL-2) and to express human CD40 ligand (hCD40L). | 3 mths

SECONDARY OUTCOMES:
To determine whether MHC- restricted or unrestricted anti-tumor immune responses are induced by SC injections of B-CLL cells which have been modified ex vivo to secrete hIL-2 and to express hCD40L | 15 yrs
To obtain preliminary data on the anti-tumor effects of this treatment regimen | 15 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (1):
- The Methodist Hospital, Houston, Texas, United States